CLINICAL TRIAL: NCT03011424
Title: Early Postoperative Extracorporal Liver Support Therapy (ELS) as a Tool to Manage Post Hepatectomy Liver Failure (PLF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Lars Lundell, Professor, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/149-31/2
Record Dates: First submitted 2016-10-24; First posted 2017-01-05 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Post Hepatectomy Liver Failure
Keywords: Liver resection; post hepatectomy liver failure; liver dialysis; encephalopathy; mortality
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Early Postoperative Extracorporal Liver Support Therapy (ELS) (Experimental): Early Postoperative Extracorporal Liver Support Therapy (ELS) by using the Molecular Adsorbent Recirculating System (MARS)
  Interventions: Device: Extracorporeal liver support therapy (ELS)

INTERVENTIONS:
Device: Extracorporeal liver support therapy (ELS) — ELS by using the Molecular Adsorbent Recirculating System (MARS) is based on a modified haemodialysis that allows the removal of water-soluble and protein bound toxins over an albumin-coated high flux membrane against recycled exogenous albumin.

SUMMARY:
Early postoperative extracorporal liver support therapy (ELS) as a tool to manage post hepatectomy liver failure (PLF).

Post-operative liver failure (PLF) has been identified as a major risk factor leading to increased morbidity and mortality. The incidence of PLF varies largely between 0-30%, and may be accounted for the main reason of postoperative mortality related to liver surgery (reported figures ranging from 18 to 75 %).

Currently, there are only a few treatment options for PLF, mainly restricted to the treatment of complications like bile leakage, infections as well as the prevention of further liver damage caused by e.g. thrombosis or haemorrhage as well as administration of liver toxic drugs. Recently the international study group on liver surgery (ISGLS) published criteria for a new definition of PLF which will greatly facilitate the comparison of results from future studies on a variety of aspects on liver failure.

ELS by using the Molecular Adsorbent Recirculating System (MARS) is based on a modified haemodialysis that allows the removal of water-soluble and protein bound toxins over an albumin-coated high flux membrane against recycled exogenous albumin. Thus, MARS can support the compromised detoxification capacity of the liver as well as improve physiological parameters. This would offer the potential for temporary support for the harmed liver after liver resection allowing for a more uneventful recovery.

For obvious reasons previous reports contain few patients, present heterogonous treatment groups and all suffer from lack of standardized treatment protocols. Few if any surviving patients, thus providing no evidence to encourage ELS as a possible treatment option for patients suffering of PLF. However, studies with defined patient populations and treatments according to a predefined standardised treatment protocol are warranted.

Primary issues to be addressed:

1. Can ELS be applied in an early phase of PLF?
2. Is ELS safe and feasible for the treatment of PLF when practised according to a predefined protocol?

Secondary issues to be addressed:

1. The development of predictive laboratory-chemical markers of liver failure
2. Indirect measures of portal flow and portal pressure
3. Indocyanine green clearance (ICG) under ELS treatment
4. Clearance of toxic products as assessed in aliquots taken from the dialysate

DETAILED DESCRIPTION:
Primary issues to be addressed

1. Can ELS be applied in an early phase of PLF?
2. Is ELS safe and feasible for the treatment of PLF when practised according to a predefined protocol?

Secondary issues to be addressed

1. The development of predictive laboratory-chemical markers of liver failure
2. Indirect measures of portal flow and portal pressure
3. Indocyanine green clearance (ICG) under ELS treatment
4. Clearance of toxic products as assessed in aliquots taken from the dialysate

Design

* Prospective phase 1 safety and feasibility study

Study Population

* 10 consecutive patients being subjected to extended liver surgery (at least right sided or extended right/left sided hemihepatectomy)

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Patients subjected for major liver surgery (4 or more Couinaud segments, ca. 50 % or more of total liver volume)
* Pre-operative chemotherapy and/or biological agents are allowed
* Liver cirrhosis Child Pugh Score A is allowed

Exclusion Criteria:

* Any contra indication for ELS such as uncontrolled active bleeding or platelet counts <20.000 /µl
* Macroscopic liver cirrhosis (Child Pugh Score B and C)
* Inability or unwilling to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of PLF patients who develop serious adverse events during ELS according to SOFA scores and Westhaven criteria | First two weeks postoperatively after major hepatectomy
  At least five sessions of Mars. SOFA (score 1-4).
Number of PLF patients who develop serious adverse events during ELS | First two weeks postoperatively after major hepatectomy
  At least five sessions of Mars. Westhaven (criteria 1-4)

SECONDARY OUTCOMES:
The predictive value of liver enzymes and bilirubin changes as marker of liver failure | First two weeks postoperatively after major hepatectomy
  At least five sessions of Mars. Liver enzymes measured( liver transaminases microkat/L ), bilirubin (mmol/L)
Portal flow (ml/minute) before and during ELS | First two weeks postoperatively after major hepatectomy
  At least five sessions of Mars
To assess liver function by use of Indocyanine green clearance (ICG)(% clearance/unit time) under ELS treatment | First two weeks postoperatively after major hepatectomy
  At least five sessions of Mars
Portal pressure (cmH2O) before and during ELS | First two weeks postoperatively after major hepatectomy
  At least five sessions of Mars

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Isaksson, Ass prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Surgery Gastrocentrum Karolinska Univeristy Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Publication in peer reviewed journal

REFERENCES:
- [Derived] Gilg S, Sparrelid E, Engstrand J, Baumgartner R, Nowak G, Stal P, D'Souza M, Jansson A, Isaksson B, Jonas E, Stromberg C. Molecular adsorbent recirculating system treatment in patients with post-hepatectomy liver failure: Long-term results of a pilot study. Scand J Surg. 2022 Sep;111(3):48-55. doi: 10.1177/14574969221112224. Epub 2022 Aug 24. PMID 36000747